CLINICAL TRIAL: NCT02053259
Title: Walking Intervention Through Texting Study: A Factorial Trial
Brief Title: A Walking Intervention Through Text Messaging
Acronym: WalkIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Marc Adams, PhD, MPH, Associate Professor, College of Health Solutions, Arizona State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: ASU-SNHP01
Record Dates: First submitted 2014-01-31; First posted 2014-02-03 (Estimated); Results first posted 2020-07-29 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-08

CONDITIONS: Physical Activity; Behavior; Overweight; Motor Activity
MeSH Terms: conditions — Motor Activity; Behavior; Overweight | interventions — Reinforcement Machine Learning

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Adaptive Goals with Immediate Reinforcement (Experimental): Adaptive Physical Activity Goals, Immediate Financial Reinforcement
  Interventions: Behavioral: Adaptive Goals; Behavioral: Reinforcement
- Adaptive Goals with Delayed Reinforcement (Experimental): Adaptive Physical Activity Goals, Delayed Financial Reinforcement
  Interventions: Behavioral: Adaptive Goals
- Static Goals with Immediate Reinforcement (Experimental): Static Physical Activity Goals, Immediate Financial Reinforcement
  Interventions: Behavioral: Reinforcement; Behavioral: Static Goals
- Static Goals with Delayed Reinforcement (Active Comparator): Static Physical Activity Goals, Delayed Financial Reinforcement
  Interventions: Behavioral: Static Goals

INTERVENTIONS:
Behavioral: Adaptive Goals
  Arms: Adaptive Goals with Delayed Reinforcement; Adaptive Goals with Immediate Reinforcement
Behavioral: Reinforcement
  Arms: Adaptive Goals with Immediate Reinforcement; Static Goals with Immediate Reinforcement
Behavioral: Static Goals
  Arms: Static Goals with Delayed Reinforcement; Static Goals with Immediate Reinforcement

SUMMARY:
The purpose of this study is to develop and evaluate adaptive goal setting and feedback interventions (Adaptive Interventions) to promote physical activity behaviors and compare it to static physical activity interventions (Static Interventions) using two levels of goal setting (Adaptive Goals vs. Static Goals) and two levels of reinforcement procedures (Praise/Rewards and No Praise/Rewards) in a 2 x 2 factorial randomized controlled trial. All four groups will receive the intervention via a semi-automated text message system developed by the investigators study team.

The primary aim of this study will be to:

1. Evaluate whether the adaptive interventions result in greater change in physical activity (pedometer-measured steps/day) compared to the static Intervention groups. HYPOTHESES: Participants in the adaptive interventions will increase their steps/day more than participants in the Static Intervention groups. The Adaptive Goals and Reinforcement Group will outperform the other 3 groups.

   The secondary aims of this study will be to:
2. Evaluate the effectiveness of the adaptive and static goal interventions in improving anthropometric, cardiovascular fitness, and cardiometabolic risk factors. HYPOTHESES: Participants in the adaptive interventions will show greater improvements in fitness, lean and fat body mass, and serum biomarkers than participants in the Static Intervention groups. The Adaptive Goals and Reinforcement Group will outperform the other 3 groups.
3. to assess participants' satisfaction with the overall program.

ELIGIBILITY:
Inclusion Criteria:

* women and men of all races/ethnicities living in Maricopa County, Arizona.

Exclusion Criteria:

* be between 18 and 60 years old
* currently not exceeding physical activity recommendations determined by the International Physical Activity Questionnaire (IPAQ short form).
* not have a medical condition based on the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) that requires supervised physical activity
* not taking medication(s) that would prohibit a moderate intensity physical activity program
* have a body mass index between 25 and 55 kg/m2
* not be currently pregnant or planning to become pregnant in the next 4 months
* not be planning to leave Maricopa County for 10 days or more in the next 4 months
* not planning to move from Maricopa County in the next 4 months
* not currently in another physical activity, diet, or weight loss program (e.g. weight watchers)
* have access to Microsoft Windows (XP, Vista, 7, 8) or Mac (10.5+) operating systems on computer with a USB port on a daily basis
* have daily access to email and the internet
* have a mobile phone with text messaging capabilities and be willing to send and receive up to 3-5 text messages per day.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State Univertsity, School of Nutrition and Health Promotion, Phoenix, Arizona, United States

REFERENCES:
- [Background] Hurley JC, Hollingshead KE, Todd M, Jarrett CL, Tucker WJ, Angadi SS, Adams MA. The Walking Interventions Through Texting (WalkIT) Trial: Rationale, Design, and Protocol for a Factorial Randomized Controlled Trial of Adaptive Interventions for Overweight and Obese, Inactive Adults. JMIR Res Protoc. 2015 Sep 11;4(3):e108. doi: 10.2196/resprot.4856. PMID 26362511
- [Result] Adams MA, Hurley JC, Todd M, Bhuiyan N, Jarrett CL, Tucker WJ, Hollingshead KE, Angadi SS. Adaptive goal setting and financial incentives: a 2 x 2 factorial randomized controlled trial to increase adults' physical activity. BMC Public Health. 2017 Mar 29;17(1):286. doi: 10.1186/s12889-017-4197-8. PMID 28356097
- [Result] Phillips CB, Hurley JC, Angadi SS, Todd M, Berardi V, Hovell MF, Adams MA. Delay Discount Rate Moderates a Physical Activity Intervention Testing Immediate Rewards. Behav Med. 2020 Apr-Jun;46(2):142-152. doi: 10.1080/08964289.2019.1570071. Epub 2019 Apr 11. PMID 30973315

RESULTS

PARTICIPANT FLOW:
Groups:
- Adaptive Physical Activity Goals With Immediate Reinforcement: Adaptive Physical Activity Goals with Immediate Reinforcement
- Adaptive Physical Activity Goals With Delayed Reinforcement: Adaptive Physical Activity Goals with Delayed Reinforcement
- Static Physical Activity Goals With Immediate Reinforcement: Static Physical Activity Goals with Immediate Reinforcement
- Static Physical Activity Goals With Delayed Reinforcement: Static Physical Activity Goals with Delayed Reinforcement
Period: Overall Study
Arm/Group | Adaptive Physical Activity Goals With Immediate Reinforcement | Adaptive Physical Activity Goals With Delayed Reinforcement | Static Physical Activity Goals With Immediate Reinforcement | Static Physical Activity Goals With Delayed Reinforcement
Started | 25 | 24 | 24 | 23
Completed | 25 | 24 | 24 | 23
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Adaptive with Immediate Rewards
- Arm 2: Adaptive with Delayed Rewards
- Arm 3: Static with Immediate Rewards
- Arm 4: Static with Delayed Non-Contingent Rewards
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Total
Number analyzed (Participants) | 25 | 24 | 24 | 23 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (10.16) | 44.5 (10.70) | 38.4 (8.22) | 40.3 (7.91) | 41.0 (9.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 17 | 19 | 16 | 74
  Male | 3 | 7 | 5 | 7 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 6 | 3 | 19
  Not Hispanic or Latino | 19 | 20 | 18 | 20 | 77
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 24 | 23 | 96

OUTCOME MEASURES:

1. Primary Outcome: Change in Fitbit-measured Steps/Day and Moderate-to-vigorous Physical Activity Between Study Arms.
Description: Given this study used a 2 condition (adaptive vs. static goals) x 2 condition (immediate vs. delayed financial reinforcement) randomized factorial design we report main effects for each condition. Sample sizes for main effects will be 96 participants for each comparison (Adaptive vs. Static goals or Immediate vs. Delayed Reinforcement) as the other condition. Consistent with proper analyses of factorial designs, main effects for the goal setting conditions pool participants across reinforcement conditions, and main effects for reinforcement conditions pool participants across goal setting conditions.
Time Frame: Daily for 4 months
Population: 2x2 factorial design main effects reported. Main effects for goal setting (n=49 for adaptive vs. n=47 for static) and reinforcement conditions (n=49 for immediate reinforcement vs. n=47 for delayed, non-contingent reinforcement).
Measure: Mean (Standard Deviation); unit: steps
Groups:
- Adaptive Goals: Adaptive goals
- Static Goals: Static goals
- Immediate Reinforcement: Immediate reinforcement
- Delayed Non-contingent Reinforcement: Delayed non-contingent reinforcement
Arm/Group | Adaptive Goals | Static Goals | Immediate Reinforcement | Delayed Non-contingent Reinforcement
Number analyzed (Participants) | 49 | 47 | 49 | 47
steps | 9695 (3948) | 9836 (3930) | 10562 (4032) | 8969 (3802)

2. Secondary Outcome: Change in Fitness (VO2max) Between Study Arms.
Time Frame: Baseline and 4 months
Reporting Status: Not Posted, anticipated posting 2023-01

3. Secondary Outcome: Changes in Body Mass Index and Body Composition Measured by Dual-energy X-Ray Absorptiometry (DEXA) Between Study Arms.
Time Frame: Baseline and 4 months
Reporting Status: Not Posted, anticipated posting 2023-01

4. Secondary Outcome: Changes to iAortic Pulse Wave Velocity Assessed With the SphymocorTM Between Study Arms.
Time Frame: Baseline and 4 months
Reporting Status: Not Posted, anticipated posting 2023-01

5. Secondary Outcome: Changes to Cardiovascular-disease (CVD) Risk and Inflammatory Markers (e.g. Glucose, Insulin, Lipids, Adhesion Molecules and Hemostatic Factors) Between Groups.
Time Frame: Baseline and 4 months
Reporting Status: Not Posted, anticipated posting 2023-01

6. Secondary Outcome: Changes to Self-reported Physical Activity Measured by the International Physical Activity Questionnaire (IPAQ).
Time Frame: Baseline and 4 months
Reporting Status: Not Posted, anticipated posting 2023-01

ADVERSE EVENTS:
Time Frame: Continuously over the course of the 4-month intervention period.
Groups:
- Arm 1: Adaptive Goals, Reinforcement
  Adaptive Goals
  Reinforcement
- Arm 2: Adaptive Goals, No Reinforcement
  Adaptive Goals
- Arm 3: Static Goals, Reinforcement
  Reinforcement
  Static Goals
- Arm 4: Static Goals, No reinforcement
  Static Goals
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24 | 0/24 | 0/23

LIMITATIONS AND CAVEATS:
Not all of the secondary outcome data have been analyzed and some results are pending review by a journal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes